CLINICAL TRIAL: NCT05265793
Title: A Multicenter, Open, Single Arm, Phase II Clinical Study of Camrelizumab Combined With Apatinib in the Treatment of Advanced Sarcomatoid Carcinoma or Carcinosarcoma
Brief Title: Camrelizumab Combined With Apatinib in the Treatment of Advanced Sarcomatoid Carcinoma or Carcinosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDCC-SC-001
Record Dates: First submitted 2021-11-23; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: PD-1 Immunotherapy; VEGFR-TKI; Sarcomatoid Carcinoma; Carcinosarcoma
MeSH Terms: conditions — Carcinoma; Carcinosarcoma | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: Regimen: Apatinib: 250mg qd, po, 4 weeks as a cycle, continuous medication until disease progression, death or intolerable toxicity; Carrelizumab: administered intravenously with a fixed dose of 200mg, administered intravenously (without preventive medication), each infusion for 30min (no less than 20min, no more than 60min), administered once every two weeks until disease progression, death or intolerable toxicity. The maximum period is 2 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab Combined With Apatinib (Experimental): Apatinib tablets: 250mg qd.po, 4 weeks as a cycle, continuous medication until disease progression, death or intolerable toxicity;
  Camrelizumab: administered intravenously with a fixed dose of 200mg, administered intravenously (without preventive medication), each infusion for 30min (no less than 20min, no more than 60min), administered once every two weeks until disease progression, death or intolerable toxicity. The maximum period is 2 years.
  The curative effect was evaluated every 8 weeks.
  Interventions: Drug: Camrelizumab Combined With Apatinib

INTERVENTIONS:
Drug: Camrelizumab Combined With Apatinib — After signing the informed consent, the selected patients received Camrelizumab combined with Apatinib. Treatment until disease progression and intolerable adverse reactions occur
  Other Names: PD-1 immunotherapy and VEGFR-TKIs

SUMMARY:
This study is to explore the treatment of advanced sarcomatoid carcinoma or Carcinosarcoma with Carrelizumab combined with Apatinib, in order to provide guidance and experience for new combined therapy in clinic.

DETAILED DESCRIPTION:
A number of clinical studies have shown that PD-1 immunotherapy combined with anti-vascular target drugs has achieved good clinical efficacy in primary liver cancer, nasopharyngeal carcinoma, esophageal cancer and other tumors. For sarcomatoid carcinoma, which is a rare tumor with large heterogeneity, poor treatment effect and poor prognosis, clinicians are facing great confusion on how to find a good treatment regimen in clinic. The purpose of this study is to explore the treatment of advanced sarcomatoid carcinoma with PD-1 antibody Camrelizumab combined with anti-vascular target drug Apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 75 years old, and gender is not limited;
2. Advanced patients with sarcomatoid carcinoma or carcinosarcoma confirmed by histopathology;
3. Patients with sarcomatoid carcinoma who have not received systematic drug treatment or have received first-line treatment;
4. The physical condition score (PS) of Eastern cancer cooperation group (ECoG) was 0 ~ 2;
5. The expected survival time is more than 3 months;
6. Within 7 days (including 7 days) before screening, the laboratory test data shall be Calculation: neutrophil count ≥ 1.5 × 109 / L, platelet count ≥ 90 × 109 / L, hemoglobin ≥ 90g / L (no blood transfusion within 14 days), total serum bilirubin ≤ 1.25 times the upper limit of normal (ULN); ALT and AST ≤ 2.5 x ULN (patients with liver metastasis ≤ 5x ULN); Serum creatinine ≤ 1.25 x ULN;
7. Measurable lesions (RECIST 1.1 standard);
8. The subjects (or their legal representative / Guardian) must sign the informed consent form, indicating that they understand the purpose of the study, understand the necessary procedures of the study, and are willing to participate in the study.

Exclusion criteria

Those who have one or more of the following are not eligible for this study:

1. Patients who have previously received anti-vascular targeted drugs or PD-1 mAb;
2. Received any experimental drugs or antitumor drugs within 4 weeks before enrollment; History of other tumors in the past five years, except cured cervical cancer or skin basal cell carcinoma;
3. Symptomatic brain or meningeal metastasis (unless the patient has received treatment for > 6 months, the imaging result is negative within 4 weeks before entering the study, and the clinical symptoms related to the tumor are stable at the time of entering the study);
4. Clinically significant active bleeding;
5. Pregnant or lactating women; Those who are fertile and do not take adequate contraceptive measures;
6. Alcohol or drug addiction;
7. Patients with active or history of autoimmune diseases that may recur (such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulitis, etc.), or patients with high risk (such as organ transplantation and immunosuppressive treatment). Except for autoimmune hypothyroidism requiring hormone replacement therapy only or skin diseases without systemic treatment.
8. Patients requiring systemic corticosteroids (equivalent to > 10mg prednisone / day) or other immunosuppressive drugs within 14 days before enrollment or during the study. Use topical or inhaled glucocorticoids, or use glucocorticoids for short-term (≤ 7 days) to prevent or treat non autoimmune and infrequent allergic diseases.
9. Important organ failure or other serious diseases, including interstitial pneumonia, clinically related coronary artery disease, cardiovascular disease, or myocardial infarction, congestive heart failure, unstable angina pectoris, symptomatic pericardial effusion or unstable arrhythmia within 6 months before enrollment;
10. Have a history of infection with human immunodeficiency virus, or suffer from other acquired and congenital immunodeficiency diseases, or have a history of organ transplantation or stem cell transplantation;
11. Patients with chronic hepatitis B or active hepatitis C. HBV carriers, stable hepatitis B after treatment (DNA titer less than 103 copies /ml) and cured hepatitis C patients (negative for HCV RNA test) can be enrolled.
12. Serious neurological or psychiatric history; Severe infection; Active disseminated intravascular coagulation or other concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study according to the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-11-21 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | the rate of patients with CR and PR, through study completion, an average of 1 year
  objective response rate

SECONDARY OUTCOMES:
OS | from the time signing of ICF until the date of death from any cause, assessed up to 36 months
  overall survival
PFS | from the time signing of ICF until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  progression free survival
AE | the adverse events rate and types of all enrolled patients, through study completion, an average of 1 year
  the adverse events of all enrolled patients
DCR | the rate of patients with CR, PR and SD, through study completion, an average of 1 year
  disease control rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided